CLINICAL TRIAL: NCT05735327
Title: Effectiveness and Safety of Brigatinib Treatment as First-line Therapy Administered to ALK Positive Non-Small Cell Lung Cancer (NSCLC) Patients. Prospective, Multicenter, Observational Study
Brief Title: A Study of Brigatinib as Preferred First Therapy for Adults With Non-Small Cell Lung Cancer (NSCLC) ENTIRETY
Acronym: ENTIRETY
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Brigatinib-4004
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Drug Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimen collected would be blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brigatinib: Participants receiving Brigatinib as part of their first-line treatment in scope of their routine clinical practice within the frames of National Drug Program (NDP) will be observed at baseline, and every 3 months (± 1 month) at routine follow-up for up to 33 months.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — As this is an observational study, no intervention will be administered.

SUMMARY:
This is a study of brigatinib in adults with Non-Small Cell Lung Cancer (NSCLC). The main aim of this study is to learn about the time period in which the condition does not worsen after the participant has received brigatinib. Another aim is to learn about the overall rate of participants who respond to the treatment with brigatinib.

Participants will receive brigatinib as part of their normal clinical practice. Data will be collected during regular visits to the hospital (a total of up to 12 visits is planned throughout study duration).

DETAILED DESCRIPTION:
This is a non-interventional, prospective study of Polish participants with ALK positive NSCLC receiving Brigatinib as their first line of treatment in the scope of routine clinical practice within the frames of National Drug Program (NDP). This study will evaluate progression-free survival (from the time of the first dose of brigatinib).

This study will enrol approximately 50 participants. Participants will be enrolled in the following cohort to be observed at baseline, and every 3 months up to 33 months:

• Brigatinib

This multi-center trial will be conducted in Poland. The overall duration of the study will include approximately 18 months of enrolment and approximately 33 months of data collection and follow-up.

ELIGIBILITY:
Inclusion Criteria

1. Adult (aged ≥18) ALK positive NSCLC participants receiving brigatinib as a first-line treatment in the scope of NDP.
2. Participants willing to participate in the study and signed ICF.

Exclusion Criteria

1. Current or planned participation in an interventional clinical trial for ALK positive non-small cell lung cancer (NSCLC).
2. Cognitive incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with ALK positive NSCLC who received brigatinib in first-line treatment in Poland.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Real-World Progression Free Survival (rwPFS) | Up to 33 months
  rwPFS is defined as the time from starting treatment to the time of radiographic progression according to Response evaluation criteria in solid tumors (RECIST) v1.1 criteria.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 33 months
  OS is defined as the time from starting treatment with brigatinib until death due to any cause or loss to follow-up.
Real-World Overall Response Rate (rwORR) | Up to 33 months
  rwORR (including intracranial response) is defined as the sum of the partial and complete response according to RECIST version 1.1. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Complete response is defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm.
Time to Discontinuation (TTD) | Up to 33 months
  TTD is defined as the time from starting treatment to the time to treatment discontinuation due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (12):
- Poland (12):
  - Dolnoslskie Centrum Onkologii, Pulmonologii i Hematologii, Wroclaw, Dolnoslskie
  - Szpital Kliniczny im. Heliodora Swiecickiego UM wPoznaniu., Poznan, Greater Poland Voivodeship
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii w Poznaniu, Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im.Prof. F. Lukaszczyka w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie- Panstwowy Instytut Badawczy Oddzial w Krakowie, Krakow, Lesser Poland Voivodeship
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II w Krakowie, Krakow, Lesser Poland Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin, Lublin Voivodeship
  - Instytut Gruzlicy i Chorob Pluc, Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie, Panstwowy Instytut Badawczy, Warsaw, Masovian Voivodeship
  - Podkarpackie Centrum Chorob Pluc, Rzeszów, Podkarpackie Voivodeship
  - Centrum Pulmonologii i Torakochirurgii w Bystrej, Bystra, Slskie
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 2 im. Wojskowej Akademii Medycznej Uniwersytetu Medycznego w Lodzi Centralny Szpital Weteranow, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/f64756166dc44be0?idFilter=%5B%22Brigatinib-4004%22%5D